CLINICAL TRIAL: NCT00456443
Title: Invasive Infections in Children With Hemoglobinopathies. A Clinical Descriptive Retrospective Study.
Brief Title: Invasive Infections in Children With Hemoglobinopathies
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Other Study IDs: 4140905.EMC
Record Dates: First submitted 2007-04-04; First posted 2007-04-05 (Estimated); Last update posted 2007-04-05 (Estimated); Status verified 2007-04

CONDITIONS: Thalassemia; Sickle Cell Anemia
Keywords: Thalassemia; Sickle cell anemia; Splenectomy; Infections; Streptococcal Pneumonia
MeSH Terms: conditions — Thalassemia; Anemia, Sickle Cell; Infections; Pneumonia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Historical records

SUMMARY:
Patients diagnosed as having hemoglobinopathies are exposed to serious bacterial infections, principally those patients that underwent splenectomy. Since the introduction of anti pneumococcal vaccine the incidence decreased significantly but other bacteria besides encapsulated bacteria takes place as principal cause of invasive infections. The purpose of this study is to analyse in a retrospective study the incidence of those infections in a group of patients suffering from thalassemia and sickle cell anemia treated in our clinic.

ELIGIBILITY:
Inclusion Criteria:

* All patients treated in the Pediatric Hematology Unit.

Max Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200
Dates: Start 2006-01; Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Koren, MD, Study Director — Pediatric Hematology Unit, Ha'Emek Medical Center; Waheeb Sakran, MD, Principal Investigator — Pediatric Dpt B - Ha'Emek Medical Center
Locations (1):
- Pediatric Hematology Unit and Pediatric Dpt B - HaEmek Medical Center, Afula, Israel